CLINICAL TRIAL: NCT01062685
Title: Near Infrared Spectroscopy (NIRS) to Measure Tissue Oxygen Saturation (St02)
Brief Title: Near Infrared Spectroscopy (St02)
Acronym: St02
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Hutchinson Technology Inc (Industry); Astute Medical, Inc. (Industry); Axis Shield Diagnostics Ltd (Industry)
Responsible Party: Principal Investigator, Nathan Shapiro, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2008P000323
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Septic Shock
Keywords: septic shock; sepsis; St02; Near Infrared Spectroscopy; NIRS
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Shock Cohort: The SHOCK cohort will meet the American College of Chest physicians/Society of Critical Care Medicine criteria for septic shock, specifically:
  * 1) Suspected infection
  * 2) Any two of four criteria of systemic inflammatory response:
    * a. Temperature > 100.4° or < 96.8° F
    * b. Heart rate > 90 beats/minute
    * c. Respiratory rate > 20 breaths/min. or PaCO2 < 32 mm Hg
    * d. WBC >12,000 or < 4000 cells/µL or > 10% bands
  * 3) Hypotension despite adequate fluid resuscitation:
    * a. SBP < 90 mm Hg after 20cc/kg crystalloid
  Interventions: Diagnostic Test: Near-infrared spectroscopy assessment
- Sepsis cohort: The SEPSIS cohort will to meet:
  * 1) Suspected infection
  * 2) Any two of four criteria of systemic inflammatory response:
    * a. Temperature > 100.4° or < 96.8° F
    * b. Heart rate > 90 beats/minute
    * c. Respiratory rate > 20 breaths/min. or PaCO2 < 32 mm Hg
    * d. WBC >12,000 or < 4000 cells/µL or > 10% bands
  * 3) Absence of refractory hypotension
  Interventions: Diagnostic Test: Near-infrared spectroscopy assessment
- Non-Infected controls: The third cohort will be comprised of uninfected ED control patients who met the criteria of no suspected infection, no SIRS criteria met and no evidence of hypoperfusion that are age and sex matched on a 1:1 basis with the shock cohort.
  Interventions: Diagnostic Test: Near-infrared spectroscopy assessment

INTERVENTIONS:
Diagnostic Test: Near-infrared spectroscopy assessment — The InSpectra StO2 Tissue Oxygenation Monitor (model 650; Hutchinson Technology, Hutchinson, MN, USA) with probes spaced at 15 mm will be utilized to obtain StO2 measurements.
  Following a minimum initial five-minute stabilization period, the initial StO2 will be measurement and then a Vasoocclusive Testing Procedure (VOT) will be performed using an automated tourniquet (Delfi Tourniquet System; Delfi Medical Innovations, Inc, Vancouver, BC, Canada), insufflated to 50 mmHg over the patient's SBP for a period of three minutes.
  Other Names: NIRS assessment

SUMMARY:
The overall hypotheses of this project is that Near Infrared Spectroscopy (NIRS) can be used to identify morbidity, mortality, and resource utilization in patients with sepsis and septic shock.

DETAILED DESCRIPTION:
Near-infrared spectroscopy (NIRS) noninvasively measures peripheral tissue oxygen saturation (StO2), offering promise as a guide in the early treatment of severe sepsis; however, the role and utility of this technology is still evolving.

There are three main NIRS measurements reported in the literature: continuous StO2 measurement (StO2 initial), StO2 occlusion slope (StO2 downslope) in response to VOT testing and StO2 recovery slope (StO2 upslope) in response to vasoocclusive testing. The purpose of this study is to assesses the association of each of these parameters with severity of illness, organ dysfunction and death.

This study will utilize the Hutchinson InSpectra StO2 tissue oxygenation monitor, which is FDA approved for use in monitoring patients during circulatory or perfusion examinations of skeletal muscle, or when there is a suspicion of compromised circulation.

ELIGIBILITY:
There will be three cohorts enrolled in this study: (1) Septic Shock, (2) Sepsis and (3) Controls.

Inclusion Criteria:

Listed on the Cohorts description.

Exclusion Criteria:

All patient cohorts will share common set of exclusion criteria:

* Age < 18 years
* Pregnancy
* Established "Do Not Resuscitate" orders prior to enrollment
* Primary diagnosis of:

  * Acute traumatic or burn injury
  * Acute cerebrovascular event
  * Acute coronary syndrome
  * Acute pulmonary edema
  * Cardiac dysrhythmia
  * Acute and active gastrointestinal bleeding
  * Acute drug overdose
  * Requirement for immediate surgery
  * Inability to obtain written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department (ED) of one of three large, urban, tertiary care facilities.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Organ Dysfunction and Severity of Illness | time 0 - 24 hrs

SECONDARY OUTCOMES:
Mortality | In hospital

CONTACTS AND LOCATIONS:
Overall Officials: Nathan I Shapiro, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Skibsted S, Arnold R, Sherwin R, Singh S, Lundy D, Nelson T, Puskarich MA, Trzeciak S, Jones AE, Shapiro NI. The association of near infrared spectroscopy-derived StO2 measurements and biomarkers of endothelial activation in sepsis. Intern Emerg Med. 2013 Sep;8(6):529-36. doi: 10.1007/s11739-013-0973-3. Epub 2013 Jul 4. PMID 23824446
- [Result] Shapiro NI, Arnold R, Sherwin R, O'Connor J, Najarro G, Singh S, Lundy D, Nelson T, Trzeciak SW, Jones AE; Emergency Medicine Shock Research Network (EMShockNet). The association of near-infrared spectroscopy-derived tissue oxygenation measurements with sepsis syndromes, organ dysfunction and mortality in emergency department patients with sepsis. Crit Care. 2011;15(5):R223. doi: 10.1186/cc10463. Epub 2011 Sep 22. PMID 21939529